CLINICAL TRIAL: NCT03363503
Title: Comparison of Efficacy and Safety of Salmeterol/Fluticasone 50/500 mcg Inhalation Powder Treatment Administered Via Capsair and Original Product Seretide Diskus 500 mcg Inhalation Powder Treatment in Patients With Moderate-severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Salmeterol/Fluticasone 50/500 mcg Inhalation Powder Via Capsair vs Seretide Diskus 500 mcg Inhalation Powder in Patients With COPD
Acronym: COPD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Adequate number of patients could not be reached in the relevant centers.
Sponsor: Neutec Ar-Ge San ve Tic A.Ş (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEU-11.15
Record Dates: First submitted 2017-11-17; First posted 2017-12-06 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: COPD
Keywords: COPD; Salmeterol/Fluticasone; Discair; Diskus; Spirometry
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Salmeterol Xinafoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salmeterol/Fluticasone Capsair® (Experimental): Salmeterol/Fluticasone 50/500 mcg Inhalation Powder (1 puff) twice daily (approximately every 12 hr) via Capsair® for 8 weeks
  Interventions: Drug: Salmeterol/Fluticasone Capsair®
- Salmeterol/Fluticasone Diskus® (Active Comparator): Salmeterol/Fluticasone 50/500 mcg Inhalation Powder (1 puff) twice daily (approximately every 12 hr) via Diskus® for 8 weeks
  Interventions: Drug: Salmeterol/Fluticasone Diskus®

INTERVENTIONS:
Drug: Salmeterol/Fluticasone Capsair® — Salmeterol/Fluticasone 50/500 mcg Inhalation Powder (1 puff) twice daily (approximately every 12 hr) via Capsair® for 8 weeks
  Other Names: Serair 50/500 mcg Capsair® Inhalation Powder
  Arms: Salmeterol/Fluticasone Capsair®
Drug: Salmeterol/Fluticasone Diskus® — Salmeterol/Fluticasone 50/500 mcg Inhalation Powder (1 puff) twice daily (approximately every 12 hr) via Diskus® for 8 weeks
  Other Names: Seretide Diskus® 500 mcg Inhalation Powder
  Arms: Salmeterol/Fluticasone Diskus®

SUMMARY:
The aim of the current study is to compare the efficacy and safety of Salmeterol/Fluticasone 50/500 mcg Inhalation Powder treatment administered via Capsair twice daily and original product Seretide Diskus 500 mcg Inhalation Powder treatment twice daily in patients with moderate-severe COPD.

Spirometric measurements will be performed at 12 different time points at pre-treatment and post-treatment (5. min, 15. min, 30. min, 1. hr, 2. hr, 3.hr, 4.hr, 6.hr, 8.hr, 10.hr and 12.hr) during the treatment visits of 11-weeks study period.

DETAILED DESCRIPTION:
The aim of the current study is to compare the efficacy and safety of Salmeterol/Fluticasone 50/500 mcg Inhalation Powder treatment administered via Capsair twice daily and original product Seretide Diskus 500 mcg Inhalation Powder treatment twice daily in patients with moderate-severe COPD.

Patients who met all the inclusion criteria will enter a 1-week run-in period with the length determine by the specific medication, during which their usual treatment will be stopped and they will receive salbutamol as required.

Following run-in period, patients will be randomly assigned to receive Salmeterol/Fluticasone 50/500 mcg as dry powder capsule for inhalation by Capsair or Salmeterol/Fluticasone 50/500 mcg as dry powder for inhalation by Diskus twice daily for 8-weeks treatment period.

Patients will be evaluated at 6 consecutive visits: baseline (enrollment), screening, treatment (treatment initiation, after 4 and 8 weeks of treatment) and after treatment (will carry out by telephone two weeks following the last dose of study medication).

Spirometric measurements will be performed at 12 different time points at pre-treatment and post-treatment (5. min, 15. min, 30. min, 1. hr, 2. hr, 3.hr, 4.hr, 6.hr, 8.hr, 10.hr and 12.hr) during the treatment visits of 11-weeks study period.

Safety will be assessed through vital signs, adverse events, serious adverse events and all cause mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥40 years with moderate-severe COPD diagnosis according to the GOLD (The Global Initiative for Chronic Obstructive Lung Disease) strategy
* Patients who have symptomatic stable moderate to severe COPD diagnosis with post-bronchodilator FEV1/ Forced Vital Capacity (FVC) <0.70, and FEV1 ≥30% and <80% of predicted normal value at screening visit
* Current smokers or ex-smokers with a smoking history of at least 10 pack-years
* Patients who have no exacerbation within last 4 weeks
* Females patients with childbearing potential using effective birth control method
* Patients whose medication unchanged within least 4 weeks
* Patients who has a capability of communicate with investigator
* Patients who accept to comply with the requirements of the protocol
* Patients who signed written informed consent prior to participation

Exclusion Criteria:

* History of hypersensitivity to long acting beta-2 agonists or corticosteroids
* History of asthma or significant chronic respiratory diseases (e.g., interstitial lung diseases, significant bronchiectasis, etc.)
* Patients who had COPD exacerbation or lower respiratory track infections that required antibiotic, oral or parenteral corticosteroid treatment within 4 weeks prior to screening visit or during run-in period
* Use of immunosupresants or systemic corticosteroids within least 4 weeks
* History of severe cardiac arrhythmia or myocardial infarction within less than 6 months
* Significant or uncontrolled disease that may preclude participant from participating in the study
* Diognosis of cancer
* History of lung volume reduction operation
* Patients vaccinated with live attenuated vaccines within 2 weeks prior to screening visit or during run-in period
* Women patients who are pregnant or nursing
* History of allergic rhinitis and atopy

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2022-04-13 (Actual); Study Completion 2022-04-13 (Actual)

PRIMARY OUTCOMES:
Mean maximum change (ml) from baseline in Forced Expiratory Volume in One Second (FEV1) | 8-weeks treatment period after randomization
  Spirometric measurements will be performed at 12 different time points at pre-treatment and post-treatment (5. min, 15. min, 30. min, 1. hr, 2. hr, 3.hr, 4.hr, 6.hr, 8.hr, 10.hr and 12.hr) during the treatment visits.
Mean percentage (%) change from baseline in | 8-weeks treatment period after randomization
  Spirometric measurements will be performed at 12 different time points at pre-treatment and post-treatment (5. min, 15. min, 30. min, 1. hr, 2. hr, 3.hr, 4.hr, 6.hr, 8.hr, 10.hr and 12.hr) during the treatment visits.
Comparison of FEV1 values at pre-dose and 2 hours post-dose | 8-weeks treatment period after randomization
  Spirometric measurement will be performed at pre-dose and 2 hours post-dose
FEV1 (AUC0-12) response [AUC: area under the curve; response defined as change from baseline] | 8-weeks treatment period after randomization
  Spirometric measurements will be performed at 12 different time points at pre-treatment and post-treatment (5. min, 15. min, 30. min, 1. hr, 2. hr, 3.hr, 4.hr, 6.hr, 8.hr, 10.hr and 12.hr) during the treatment visits.
FVC (AUC0-12) response | 8-weeks treatment period after randomization
  Spirometric measurements will be performed at 12 different time points at pre-treatment and post-treatment (5. min, 15. min, 30. min, 1. hr, 2. hr, 3.hr, 4.hr, 6.hr, 8.hr, 10.hr and 12.hr) during the treatment visits.
FEV1 (AUC12-24) response | 8-weeks treatment period after randomization
  Spirometric measurements will be performed at 12 different time points at pre-treatment and post-treatment (5. min, 15. min, 30. min, 1. hr, 2. hr, 3.hr, 4.hr, 6.hr, 8.hr, 10.hr and 12.hr) during the treatment visits.
FVC (AUC12-24) response | 8-weeks treatment period after randomization
  Spirometric measurements will be performed at 12 different time points at pre-treatment and post-treatment (5. min, 15. min, 30. min, 1. hr, 2. hr, 3.hr, 4.hr, 6.hr, 8.hr, 10.hr and 12.hr) during the treatment visits.
FEV1 (AUC0-24) response | 8-weeks treatment period after randomization
  Spirometric measurements will be performed at 12 different time points at pre-treatment and post-treatment (5. min, 15. min, 30. min, 1. hr, 2. hr, 3.hr, 4.hr, 6.hr, 8.hr, 10.hr and 12.hr) during the treatment visits.
FVC (AUC0-24) response | 8-weeks treatment period after randomization
  Spirometric measurements will be performed at 12 different time points at pre-treatment and post-treatment (5. min, 15. min, 30. min, 1. hr, 2. hr, 3.hr, 4.hr, 6.hr, 8.hr, 10.hr and 12.hr) during the treatment visits.

SECONDARY OUTCOMES:
Mean change from baseline in transition dyspnea index (TDI) after 8-weeks treatment | 8-weeks treatment period after randomization
  Transition Dyspnea Index (TDI), a measure of the degree of breathlessness, captures changes from baseline. Baseline Dyspnea Index (BDI) score is based on three domains: functional impairment, magnitude of task and magnitude of effort. BDI will be measured at day 1 prior to the first dose with domain scores ranging from 0=very severe to 4=no impairment and a total score ranging from 0 to 12(best).
Mean change from baseline in St. George's Respiratory Questionnaire (SGRQ) after 8-weeks treatment | 8-weeks treatment period after randomization
  SGRQ is a 51-item health related quality of life questionnaire and it consists of three sections; Symptoms-measuring the frequency and severity of respiratory symptoms, Activity-measuring limitation of activities by breathlessness and activities that cause breathlessness and Impacts-measuring disturbances in social and psychological functioning due to airway disease. It will be performed to evaluate quality of life of the patients by comparing pre-treatment and post-treatment values. The lowest possible value is zero and the highest 100. Higher values correspond to greater impairment in quality of life.
Mean change from baseline in symptom severity and frequency (mean change from baseline in CAT score) | 8-weeks treatment period after randomization
  The COPD Assessment Test (CAT) is a questionnaire for people with COPD. It is designed to measure the impact of COPD on a person's life, and how this changes over time. It contains 8 questions regarding symptoms with scoring rage of zero to 40 (It will be completed using a 6 point scale).
Frequency of rescue medicine (salbutamol) used | 8-weeks treatment period after randomization
  Patients will use a diary to record the daily number of puffs of rescue medication used to treat COPD symptoms.
Time to onset of bronchodilator effect and maximum effect | 8-weeks treatment period after randomization
  Spirometric measurements will be performed at 12 different time points at pre-treatment and post-treatment (5. min, 15. min, 30. min, 1. hr, 2. hr, 3.hr, 4.hr, 6.hr, 8.hr, 10.hr and 12.hr) during the treatment visits.
Adverse events, serious adverse events and all cause mortality. | 10 weeks after randomization
  Safety will be assessed through the vital signs, number of adverse events, serious adverse events and all cause mortality.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Akdeniz University Faculty of Medicine, Chest Diseases Department, Antalya
  - Republic of Turkey Ministry of Health Antalya Training and Research Hospital, Antalya